CLINICAL TRIAL: NCT01549314
Title: Cystic Fibrosis Related Bone Disease: the Role of CFTR
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Melissa Susan Putman, Assistant Professor, Massachusetts General Hospital
Other Study IDs: MGH 2012P000269
Record Dates: First submitted 2012-03-02; First posted 2012-03-09 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis Related Bone Disease
Keywords: Cystic fibrosis related bone disease; Cystic fibrosis; Ivacaftor
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Subjects with CF taking ivacaftor: Subjects with CF ages 6 to 75 years old who will be or have started taking ivacaftor within the previous 6 months
- Subjects with CF not taking ivacaftor: Subjects with CF ages 6 to 75 years old who will not be taking ivacaftor, matched for age, race, and gender with cohort 1
- Healthy subjects: Healthy subjects with no medical conditions known to affect bone between the ages of 6 to 75 years old, matched for age, race, and gender with cohort 2.

SUMMARY:
The purpose of this study is to determine whether ivacaftor, a recently FDA-approved CFTR potentiator, improves bone micro-architecture and strength in patients with cystic fibrosis with at least one G551D CFTR mutation.

DETAILED DESCRIPTION:
Ivacaftor, a CFTR potentiator, has recently been FDA approved for the treatment of cystic fibrosis in patients with at least one G551D CFTR mutation. Given the possible role of CFTR in bone, we hypothesize that this medication may also improve bone health in CF patients. The purpose of this study is to test this hypothesis using high resolution peripheral quantitative computed tomography, a research tool that measures bone micro-architecture and volumetric bone density and has the ability to detect small changes in bone that might otherwise be missed with standard bone imaging techniques such as bone density testing.

ELIGIBILITY:
COHORT 1

Inclusion Criteria:

* Age 6 to 75 years old
* Established diagnosis of CF with at least one abnormal G551D-CFTR allele
* Eligibility for and intent to start treatment with ivacaftor or started treatment with ivacaftor within previous 6 months

Exclusion Criteria:

* Psychiatric or mental incapacity that would preclude subject from assenting to study participation
* Current pregnancy
* History of organ transplantation
* History of Burkholderia dolosa infection

COHORT 2:

Subjects will be grouped by gender, age and race to match subjects in Cohort 1 within two years. Pubertal subjects will be matched by Tanner stage.

Inclusion Criteria:

* Age 6 to 75 years old
* Established diagnosis of CF

Exclusion Criteria:

* Psychiatric or mental incapacity that would preclude subject from assenting to study participation
* Current pregnancy
* History of organ transplantation
* History of Burkholderia dolosa infection

COHORT 3:

Subjects will be grouped by gender, age and race to match subjects in Cohort 2 within two years. Pubertal subjects will be matched by Tanner stage.

Inclusion criteria:

* Age 6 to 75 years old
* Clinically stable, deemed able to complete the screening, baseline, and scheduled study visits.

Exclusion criteria:

* History of significant cardiac, renal, pulmonary, hepatic, or malignant disease, current alcohol or illicit drug abuse, or major psychiatric disorder
* Current diagnoses known to affect bone metabolism, including cystic fibrosis, osteoporosis, amenorrhea >3 months (in menstruating women who are not taking oral contraceptives or have an IUD), hyperthyroidism, diabetes, hyperparathyroidism, Paget's disease, kidney stones, chronic inflammatory diseases, malabsorptive disorders, malnutrition, prolonged immobility, and skeletal dysplasias
* History of a non-digital fracture in the previous 6 months, history of one pathologic fracture, or greater than four total lifetime non-digital fractures
* Cumulative lifetime use of oral glucocorticoids for greater than 2 months
* Current or prior use of medications known to affect bone metabolism including hormone replacement therapy, anti-estrogens, bisphosphonates, calcitonin, fluoride, lithium, suppressive doses of levothyroxine, or anticonvulsants.
* Pregnancy
* BMI less than 18.5 or greater than 30 kg/m2 in subjects 18 years and older, or BMI less than 5th or greater than 95th percentile in subjects under the age of 18 years.
* Any medical or psychiatric condition or situation that would compromise subject safety, informed consent/assent, treatment compliance, follow-up measurements, or data quality

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with CF will be recruited from the Cystic Fibrosis Centers at Children's Hospital Boston and Massachusetts General Hospital. Healthy subjects will be a community sample recruited from nearby communities.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Finkelstein, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ramsey BW, Davies J, McElvaney NG, Tullis E, Bell SC, Drevinek P, Griese M, McKone EF, Wainwright CE, Konstan MW, Moss R, Ratjen F, Sermet-Gaudelus I, Rowe SM, Dong Q, Rodriguez S, Yen K, Ordonez C, Elborn JS; VX08-770-102 Study Group. A CFTR potentiator in patients with cystic fibrosis and the G551D mutation. N Engl J Med. 2011 Nov 3;365(18):1663-72. doi: 10.1056/NEJMoa1105185. PMID 22047557
- [Background] Accurso FJ, Rowe SM, Clancy JP, Boyle MP, Dunitz JM, Durie PR, Sagel SD, Hornick DB, Konstan MW, Donaldson SH, Moss RB, Pilewski JM, Rubenstein RC, Uluer AZ, Aitken ML, Freedman SD, Rose LM, Mayer-Hamblett N, Dong Q, Zha J, Stone AJ, Olson ER, Ordonez CL, Campbell PW, Ashlock MA, Ramsey BW. Effect of VX-770 in persons with cystic fibrosis and the G551D-CFTR mutation. N Engl J Med. 2010 Nov 18;363(21):1991-2003. doi: 10.1056/NEJMoa0909825. PMID 21083385
- [Background] MacNeil JA, Boyd SK. Accuracy of high-resolution peripheral quantitative computed tomography for measurement of bone quality. Med Eng Phys. 2007 Dec;29(10):1096-105. doi: 10.1016/j.medengphy.2006.11.002. Epub 2007 Jan 16. PMID 17229586
- [Background] Aris RM, Merkel PA, Bachrach LK, Borowitz DS, Boyle MP, Elkin SL, Guise TA, Hardin DS, Haworth CS, Holick MF, Joseph PM, O'Brien K, Tullis E, Watts NB, White TB. Guide to bone health and disease in cystic fibrosis. J Clin Endocrinol Metab. 2005 Mar;90(3):1888-96. doi: 10.1210/jc.2004-1629. Epub 2004 Dec 21. PMID 15613415
- [Background] Shead EF, Haworth CS, Condliffe AM, McKeon DJ, Scott MA, Compston JE. Cystic fibrosis transmembrane conductance regulator (CFTR) is expressed in human bone. Thorax. 2007 Jul;62(7):650-1. doi: 10.1136/thx.2006.075887. No abstract available. PMID 17600296
- [Derived] Putman MS, Greenblatt LB, Bruce M, Joseph T, Lee H, Sawicki G, Uluer A, Sicilian L, Neuringer I, Gordon CM, Bouxsein ML, Finkelstein JS. The Effects of Ivacaftor on Bone Density and Microarchitecture in Children and Adults with Cystic Fibrosis. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1248-e1261. doi: 10.1210/clinem/dgaa890. PMID 33258950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 27 subjects with CF taking ivacaftor were enrolled; however, 1 subject dropped out immediately after signing the consent form prior to any study procedures. No baseline data were obtained in this subject. Therefore, 26 subjects with CF taking ivacaftor were followed prospectively and were matched to the other 2 cohorts.
Period: Overall Study
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects
Started | 27 (1 subject signed the consent form but dropped out prior to any study procedures or data collection.) | 26 | 26
Completed | 23 | 21 | 24
Not Completed | 4 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects | Total
Number analyzed (Participants) | 26 | 26 | 26 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 11 | 33
  Between 18 and 65 years | 15 | 15 | 15 | 45
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.1 (13.1) | 22.8 (13.1) | 23.8 (13.2) | 23.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 15 | 45
  Male | 11 | 11 | 11 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 26 | 26 | 78
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 26 | 26 | 26 | 78
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 26 | 78

OUTCOME MEASURES:

1. Primary Outcome: Bone Microarchitecture and Strength Measures of the Radius and Tibia
Description: Change in cortical volumetric bone mineral density at the radius
Time Frame: Baseline and 24 months
Population: Subjects who were lost to follow up prior to the 24 month visit were not included in the analyses
Measure: Mean (Standard Deviation); unit: mgHA/cm3
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects
Number analyzed (Participants) | 23 | 21 | 24
mgHA/cm3 | 44.6 (53.9) | 40.1 (44.0) | 43.7 (53.8)
Statistical Analysis 1: Comparison: Subjects With CF Taking Ivacaftor vs Subjects With CF Not Taking Ivacaftor; Change from baseline to 24 months in cortical volumentric bone mineral density was determined and compared between subjects with CF taking ivacaftor and subjects with CF not taking ivacaftor; Test type: Superiority; p = 0.77, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With CF Not Taking Ivacaftor vs Healthy Subjects; Change from baseline to 24 months in cortical volumentric bone mineral density was determined and compared between subjects with CF not taking ivacaftor and healthy subjects; Test type: Superiority; p = 0.82, t-test, 2 sided

2. Secondary Outcome: Areal Bone Mineral Density as Measured by DXA
Description: Change in PA spine bone mineral density
Time Frame: Baseline and 24 months
Population: Subjects who were lost to follow up prior to the 24 month visit were not included in the analyses
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects
Number analyzed (Participants) | 23 | 21 | 24
g/cm2 | 0.032 (0.058) | 0.024 (0.043) | 0.029 (0.043)
Statistical Analysis 1: Comparison: Subjects With CF Taking Ivacaftor vs Subjects With CF Not Taking Ivacaftor; Change from baseline to 24 months in DXA PA spine bone mineral density was determined and compared between subjects with CF taking ivacaftor and subjects with CF not taking ivacaftor; Test type: Superiority; p = 0.64, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With CF Not Taking Ivacaftor vs Healthy Subjects; Change from baseline to 24 months in DXA PA spine bone mineral density was determined and compared between subjects with CF not taking ivacaftor and healthy subjects; Test type: Superiority; p = 0.78, t-test, 2 sided

3. Secondary Outcome: Bone Turnover Markers
Description: Change in osteocalcin
Time Frame: Baseline and 24 months
Population: Subjects who were lost to follow up prior to the 24 month visit were not included in the analyses
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects
Number analyzed (Participants) | 23 | 21 | 24
ng/ml | -5.36 (12.89) | -4.51 (16.27) | -4.5 (14.55)
Statistical Analysis 1: Comparison: Subjects With CF Taking Ivacaftor vs Subjects With CF Not Taking Ivacaftor; Change from baseline to 24 months in osteocalcin was determined and compared between subjects with CF taking ivacaftor and subjects with CF not taking ivacaftor; Test type: Superiority; p = 0.86, t-test, 2 sided
Statistical Analysis 2: Comparison: Subjects With CF Not Taking Ivacaftor vs Healthy Subjects; Change from baseline to 24 months in osteocalcin was determined and compared between subjects with CF not taking ivacaftor and healthy subjects; Test type: Superiority; p = 0.99, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Description: This was an observational study following subjects prospectively over time without an intervention. Any medications, including ivacaftor, were managed by subjects' physician. Therefore, adverse events associated with this study were related to study procedures only. One subject felt lightheaded after venipuncture, improved with food and water, and this was the only adverse event reported.
Arm/Group | Subjects With CF Taking Ivacaftor | Subjects With CF Not Taking Ivacaftor | Healthy Subjects
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 1/26 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With CF Taking Ivacaftor (N=26) | Subjects With CF Not Taking Ivacaftor (N=26) | Healthy Subjects (N=26)
Minor (Investigations) | 0 (0) | 1 (1) | 0 (0) — Lightheaded

LIMITATIONS AND CAVEATS:
This was a prospective observational multiple cohort study and not a randomized or interventional clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT01549314/Prot_SAP_000.pdf